CLINICAL TRIAL: NCT01505738
Title: The Effect of Bacterial Growth in Vascular Surgery Wounds to the Incidence of Postoperative Wound Infections
Brief Title: Bacterial Growth in Vascular Surgery Wounds
Status: Completed | Type: Observational
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, Principal investigator, North Karelia Central Hospital
Other Study IDs: NKCH-Surg-009
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Lower Limb Ischaemia; Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bacterial cultures: Bacterial samples are collected preoperatively from urine, nose and possible lower limb ischaemic wounds, perioperatively from inguinal area and wound edges, and twice postoperatively. In addition, in case of a wound infection, bacterial samples are taken for diagnosis as usual.
  Interventions: Other: bacterial samples

INTERVENTIONS:
Other: bacterial samples — bacterial samples taken

SUMMARY:
The amount and species of bacteria have been shown to have an effect in wound infections in several fields of surgery (such as gastrointestinal and orthopaedic surgery and the surgery of facial area). In vascular surgery, wound infections are a common and expensive complication. The aim of the present study is to investigate the prevalence of bacteria in vascular surgery wounds perioperatively, and determine whether is correlates with the incidence of wound infections postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* need for lower limb vascular by-pass surgery

Exclusion Criteria:

* allergic to cefuroxime
* patients refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients requiring lower limb vascular surgery due to ischaemic changes and/or lower limb aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
wound infection | 3 months
  incidence of wound infection after lower limb vascular surgery

CONTACTS AND LOCATIONS:
Locations (1):
- North Karelia Central Hospital, Clinic of Surgery, Joensuu, Finland